CLINICAL TRIAL: NCT00083135
Title: I-MIBG Escalating Dose Rapid Sequence Double Infusion Followed By Autologous Stem Cell Infusion For Refractory Neuroblastoma
Brief Title: N2000-01: Double Infusion of Iodine I 131 Metaiodobenzylguanidine Followed by Autologous Stem Cell Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Katherine K. Matthay, M.D., UCSF School of Medicine
Purpose: Treatment
Other Study IDs: CDR0000363631; P01CA081403 (NIH); N2000-01 (Other: NANT Consortium)
Record Dates: First submitted 2004-05-14; First posted 2004-05-17 (Estimated); Last update posted 2010-10-15 (Estimated); Status verified 2009-05

CONDITIONS: Neuroblastoma
Keywords: recurrent neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Filgrastim; Peripheral Blood Stem Cell Transplantation; 3-Iodobenzylguanidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: filgrastim
Procedure: autologous bone marrow transplantation
Procedure: peripheral blood stem cell transplantation
Radiation: iobenguane I 131

SUMMARY:
RATIONALE: Giving iodine I 131 metaiodobenzylguanidine (^131I-MIBG) may kill neuroblastoma cells by delivering radiation directly to the tumor. A stem cell transplant using the patient's stem cells may be able to replace blood-forming cells destroyed by radiation therapy.

PURPOSE: This phase I trial is studying the side effects and best dose of a double infusion of ^131I-MIBG followed by autologous stem cell transplantation in treating patients with refractory neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated red marrow radiation dose delivered and associated toxic effects of escalating activity of iodine I 131 metaiodobenzylguanidine (^131I-MIBG) followed by autologous hematopoietic stem cell transplantation in patients with refractory neuroblastoma.
* Determine the number of days after stem cell transplantation to achieve absolute neutrophil count ≥ 500/mm^3 for 3 days and platelet count ≥ 20,000/mm^3 for 3 days (without transfusions) in patients treated with this regimen.

Secondary

* Determine the response rate in patients treated with this regimen, based on lesions measurable by CT or MRI at study entry, patients with ^131I-MIBG scan-positive lesions only, and patients with minimal residual tumor in bone marrow who have complete response by immunocytology and morphology.
* Determine the tumor absorbed radiation dose in patients with measurable soft tissue lesions treated with this regimen.
* Correlate, if possible, TP53 mutations with response in patients with accessible bone marrow tumor treated with ^131I-MIBG.

OUTLINE: This is a dose-escalation, multicenter study.

* Iodine I 131 metaiodobenzylguanidine (131I-MIBG) therapy: Patients receive^131I-MIBG IV over 2 hours on days 0 and 14.

Cohorts of 3-6 patients receive escalating doses of ^131I-MIBG until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Stem cell transplantation therapy: Patients undergo autologous peripheral blood stem cell transplantation on day 28. Patients receive filgrastim (G-CSF) IV over 1 hour OR subcutaneously daily beginning on day 28 and continuing until blood counts recover.

Patients are followed every 3 months for 1 year and then annually thereafter.

PROJECTED ACCRUAL: A total of 9-18 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of neuroblastoma

  * Confirmed by at least 1 of the following methods:

    * Histology
    * Clumps of tumor cells in bone marrow with elevated urinary catecholamine metabolites
  * High-risk disease

    * Poor response to induction therapy OR relapse defined by any of the following:

      * No response, stable disease, or mixed response after a minimum of 3 prior courses of chemotherapy
      * More than 100 tumor cells per 10^5 nucleated cells on bone marrow immunocytology after at least 3 prior courses of chemotherapy
      * Progressive disease at any time during or after therapy
      * Patients with massive bone marrow invasion (more than 50% replacement of bone marrow by tumor cells) are allowed
* Must have positive iodine I 131 metaiodobenzylguanidine (^131I-MIBG) within the past 6 weeks or subsequent to any other prior antitumor therapy delivered within the past 6 weeks
* Must meet the following criteria for minimum number of autologous stem cells:

  * Unpurged peripheral blood stem cells (PBSC)

    * Minimum of 1,500,000/mm^3 CD34-positive cells/kg
    * Collected products must have < 1 tumor cell/100,000 normal cells by immunocytology
  * PBSC purged with immunomagnetic beads

    * Minimum of 1,000,000/mm^3 viable CD34-positive cells/kg
    * Collected products must have < 1 tumor cell/100,000 normal cells by immunocytology
  * CD34-positive selected PBSC products are not allowed
  * Patients who had PBSC collected previously with no immunocytological testing available may use those products provided bone marrow is tumor free by bilateral bone marrow aspirate AND biopsy for morphology is performed within 4 weeks before PBSC collection
  * Patients with no tumor involvement in bone marrow at diagnosis and PBSC collection before any disease progression do not require documentation of negative bone marrow morphology

PATIENT CHARACTERISTICS:

Age

* 1 to 30

Performance status

* ECOG 0-2

Life expectancy

* Less than 1 year

Hematopoietic

* Absolute neutrophil count ≥ 500/mm^3
* Platelet count ≥ 50,000/mm^3 (without transfusion)
* Hemoglobin ≥ 8 g/dL (transfusion allowed)

Hepatic

* AST and ALT ≤ 5 times normal
* Bilirubin < 2 times normal

Renal

* Creatinine ≤ 1.5 mg/dL
* Glomerular filtration rate OR 12-hour creatinine clearance ≥ 60 mL/min/1.73m^2

Cardiovascular

* Ejection fraction ≥ 55% by echocardiogram or MUGA OR
* Fractional shortening ≥ 30% OR above lower limit of normal by echocardiogram

Pulmonary

* Normal lung function
* No dyspnea at rest
* No exercise intolerance
* No oxygen requirement

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to cooperate physically and psychologically with radiation isolation
* No disease of any major organ system that would preclude study participation
* No active infection requiring antivirals, antibiotics, or antifungals
* No weight that would require exceeding a maximum total allowable dose of ^131I-MIBG

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 2 weeks since prior biologic or other non-myelosuppressive therapy

Chemotherapy

* See Disease Characteristics
* At least 2 weeks since prior chemotherapy
* More than 3 months since prior myeloablative therapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* At least 6 months since prior craniospinal, total abdominal, or whole lung radiotherapy
* At least 2 weeks since prior radiotherapy to any site
* No prior total body irradiation
* No prior radiotherapy to > 25% of bone marrow
* No prior ^131I-MIBG

Surgery

* Not specified

Other

* Recovered from all prior therapy
* Concurrent antifungal therapy allowed provided culture and biopsy are negative in suspected radiographic lesions
* Prior re-induction therapy for recurrent tumor allowed
* No concurrent antiretroviral therapy for HIV-positive patients
* No concurrent hemodialysis

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2004-03; Primary Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine K. Matthay, MD, Study Chair — University of California, San Francisco; Gregory Yanik, MD, Principal Investigator — University of Michigan Rogel Cancer Center; John M. Maris, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (7):
- United States (7):
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Children's Hospital Boston, Boston, Massachusetts
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin

REFERENCES:
- [Result] Matthay KK, Quach A, Huberty J, Franc BL, Hawkins RA, Jackson H, Groshen S, Shusterman S, Yanik G, Veatch J, Brophy P, Villablanca JG, Maris JM. Iodine-131--metaiodobenzylguanidine double infusion with autologous stem-cell rescue for neuroblastoma: a new approaches to neuroblastoma therapy phase I study. J Clin Oncol. 2009 Mar 1;27(7):1020-5. doi: 10.1200/JCO.2007.15.7628. Epub 2009 Jan 26. PMID 19171714
- [Result] Taggart DR, Han MM, Quach A, Groshen S, Ye W, Villablanca JG, Jackson HA, Mari Aparici C, Carlson D, Maris J, Hawkins R, Matthay KK. Comparison of iodine-123 metaiodobenzylguanidine (MIBG) scan and [18F]fluorodeoxyglucose positron emission tomography to evaluate response after iodine-131 MIBG therapy for relapsed neuroblastoma. J Clin Oncol. 2009 Nov 10;27(32):5343-9. doi: 10.1200/JCO.2008.20.5732. Epub 2009 Oct 5. PMID 19805691